CLINICAL TRIAL: NCT07403695
Title: Comparison Between Photobiomodulation Therapy on Nerve Repair Using Red and Infra-red Diode Lasers in Maxillofacial Region (A Randomized Clinical Trial)
Brief Title: Photobiomodulation Therapy on Nerve Repair Using Red and Infra-red Diode Lasers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mona oraby (Other)
Responsible Party: Sponsor-Investigator, mona oraby, Dr., Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00010556- 0008839
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Nerve Injury
Keywords: laser therapy; photobiomodulation; nerve injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 635 wavelength (Experimental)
  Interventions: Device: 635 wavelength
- 980 wavelength (Active Comparator)
  Interventions: Device: 980 wavelength

INTERVENTIONS:
Device: 635 wavelength — 635 wavelength laser
  Arms: 635 wavelength
Device: 980 wavelength — 980 wavelength laser
  Arms: 980 wavelength

SUMMARY:
Peripheral nerve injury is a major concern that drastically affects the patient's quality of life. Nowadays, several treatment options are available, including medical treatments, surgical intervention, and others. However, the trending photobiomodulation effect of laser therapy is attracting many dental professionals due to its promising results on nerve rehabilitation.

The study is intended to assess and compare laser photobiomodulation using red and infra-red diode lasers on the repair of nerve injury in the maxillofacial region.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged range from 20-50 years old
2. Patient suffering from nerve injury in the maxillofacial region for a period of 6 months or more without improvement.

Exclusion Criteria:

* 1- Patient had undergone micro-neurosurgery to correct neurosensory deficit.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-01-18 (Actual); Study Completion 2026-01-18 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 1,2,4,8,12 weeks
  from 1- 10
  1 means no pain 10 means worst pain

SECONDARY OUTCOMES:
clinical neurosensory test | 2,4,8,12 weeks
  from S0 to S4 S0 means worst neurosensory function S4 full recovery for neurosensory function

CONTACTS AND LOCATIONS:
Overall Officials: Mona S Oraby, Principal Investigator — Alexandria University
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No